CLINICAL TRIAL: NCT03220113
Title: Safety and Efficacy of De-Novo Algorithm and Formula in the Treatment of Patients With Intractable Chronic Craniofacial Neuralgia, or Chronic Migraine Headaches.
Brief Title: Treatment of Chronic Migraine Headaches.
Acronym: Migraine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corona Doctors Medical Clinics, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/05/1
Record Dates: First submitted 2017-07-11; First posted 2017-07-18 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2017-07

CONDITIONS: Chronic Migraine Without Aura, Intractable; Migraine With Typical Aura; Migraine Disorders
Keywords: Migraine; Craniofacial Neuralgia
MeSH Terms: conditions — Migraine with Aura; Migraine Disorders | interventions — Dexamethasone; Lidocaine

STUDY DESIGN:
Intervention Model Description: Prospective Open Label Study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dexamethasone,Lidocaine,Thiamine cohort (Experimental): Simultaneous administration of a combination of sterile dexamethasone phosphate total dose (bilaterally) of 20 mg, 4 mg/ml, Lidocaine Hydrochloride 1% 40 mg, 10 mg/ml, and Thiamine Hydrochloride 100 mg, 100 mg/ml in a single session into the accessible branches of the trigeminal nerve of the first, second, and third divisions, as well as into the greater and lesser occipital nerve. In first,patient placed in supine position then in prone position for comfortable access to injection site.
  De-Novo Treatment medication 'Dexamethasone, Lidocaine, Thiamine Cohort' prepared in single 1 milliliter volume sterile syringes, using 27 Gauge-30 Gauge needles.
  Interventions: Combination Product: Dexamethasone, Lidocaine, Thiamine cohort

INTERVENTIONS:
Combination Product: Dexamethasone, Lidocaine, Thiamine cohort — Bilateral and simultaneous administration of composition of De-Novo Treatment Cohort medication (Dexamethasone, Lidocaine, Thiamine) into the trigeminal and greater/lesser occipital nerves in one session.In children and hypersensitive individuals with needle phobia pre-treatment of skin with Lidocaine 2.5% Prilocaine 2.5% cream, and oral Alprazolam 0.25 mg (an Anxiolytic) 2 hours prior to initiation of procedure will be used.
  Other Names: De-Novo Treatment Cohort medication

SUMMARY:
The purpose of the study is assessment of the safety and efficacy of the De-Novo therapy in the treatment of craniofacial neuralgia and migraine headaches.This is an open-label study of simultaneous administration of combination of dexamethasone, lidocaine, and thiamine into the trigeminal nerve branches as well as greater and lesser occipital nerve bilaterally in one session.

Patients who meet the exclusion and inclusion criteria are eligible for trial if they have experienced chronic migraine and craniofacial pain not responding to other prior therapies.

DETAILED DESCRIPTION:
A combination of dexamethasone, lidocaine and thiamine (pat.), may bring changes in the pattern of sympathetic and parasympathetic nerve signaling at the level vasa nervorum. These changes may down-regulate the hyperexcitable sympathetic signals at the level of adventitia and consequently the medial layer of vasa nervorum and providing long term relief from migraine headaches. However, a bilateral and simultaneous treatment of trigeminal and occipital nerves in migraine and craniofacial neuralgia using a combination of dexamethasone, thiamine and lidocaine has been rarely studied.

The objective of this study is to assess the safety and efficacy of concomitant administration of dexamethasone, lidocaine, and thiamine compounds into the trigeminal nerve branches, the greater and lesser occipital nerve for the treatment of chronic migraine, and craniofacial neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* • Age: 10-90 years

  * Ability to describe headache and its symptoms
  * Ability to read, comprehend, and legibly and reliably record information
  * Ability to provide written, informed consent, and respond to pre and post treatment questionnaires, children's guardian accepts responsibility. Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures
  * Already diagnosed with chronic craniofacial neuralgia and chronic migraine headache
  * Exhausted all or most of available abortive and preventive treatment modalities.

Exclusion Criteria:

* • Uncontrollable hypertension, acute Myocardial Infarct within last 6 months

  * History of cerebral vascular aneurysm/known atherosclerosis of cerebral system, brain tumor
  * Implanted of neuro-stimulator, trigeminal tractotomy, neurectomy partial or complete, history of gamma knife treatment, microsurgical decompression procedure.
  * Hypersensitivity or allergy to any components of De-Novo formula
  * Presence or known anatomic craniofacial deformities or severe spondylosis/spondylolisthesis of cervical spine, profound dental caries, Maxillofacial deformities
  * Pregnancy and current breast feeding status
  * Headaches attribute to acute head and neck injuries, chronicity of cervicogenic headaches
  * Skin infection or micro abscesses dermatogen or dental, ongoing treatment for Methicillin Resistant Streptococcus Aureus ( MRSA) unless treatment completed.

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the safety to the De-Novo treatment formula in study patients | 5 weeks
  Study assesses the safety of the De-Novo algorithm( if patients who receive this treatment will experience any major adverse reactions due to the medication combination )within the next 5 weeks following treatment. Participants will be interviewed after the initial treatment weekly, for 5 weeks to evaluate for any possible adverse events, hospitalization, or treatment. Any significant adverse event in over 45% of participants, may project end of the trial.

SECONDARY OUTCOMES:
Assessment of the clinical response to the De-Novo treatment formula in study patients consisting of a lone composite measure | 12 months
  Assessment of the clinical response to the De-Novo treatment formula in study patients.
  Study assesses the efficacy parameters of the study ( i.e. the change in baseline frequency of migraine attack in patients post initial treatment ), and functionality status based on continuation of work performance and return to work or school.
  Therefore, the Outcome of study consisting of multiple measures and present lone composite measure.

CONTACTS AND LOCATIONS:
Overall Officials: Faro T. Owiesy, M.D., Principal Investigator — Corona Doctors Medical Clinics, Inc.
Locations (1):
- Corona Doctors Medical Clinics Inc, Corona, California, United States

IPD SHARING:
Plan to Share IPD: No
No sharing suggested at this time

REFERENCES:
- [Background] Sechi G, Serra A. Wernicke's encephalopathy: new clinical settings and recent advances in diagnosis and management. Lancet Neurol. 2007 May;6(5):442-55. doi: 10.1016/S1474-4422(07)70104-7. PMID 17434099
- [Background] Negovskii VA. [History of resuscitation in the USSR]. Vestn Akad Med Nauk SSSR. 1975;(12):26-9. No abstract available. Russian. PMID 775837
- [Background] Johri S, Shetty S, Soni A, Kumar S. Anaphylaxis from intravenous thiamine--long forgotten? Am J Emerg Med. 2000 Sep;18(5):642-3. doi: 10.1016/s0735-6757(00)90303-6. No abstract available. PMID 10999594
- [Background] Morinville V, Jeannet-Peter N, Hauser C. Anaphylaxis to parenteral thiamine (vitamin B1). Schweiz Med Wochenschr. 1998 Oct 31;128(44):1743-4. PMID 9846348
- [Background] Van Haecke P, Ramaekers D, Vanderwegen L, Boonen S. Thiamine-induced anaphylactic shock. Am J Emerg Med. 1995 May;13(3):371-2. doi: 10.1016/0735-6757(95)90221-X. No abstract available. PMID 7755837
- [Background] Wrenn KD, Murphy F, Slovis CM. A toxicity study of parenteral thiamine hydrochloride. Ann Emerg Med. 1989 Aug;18(8):867-70. doi: 10.1016/s0196-0644(89)80215-x. PMID 2757284
- [Background] De Bold JF, Ruppert PH, Clemens LG. Inhibition of estrogen-induced sexual receptivity of female hamsters: comparative effects of progesterone, dihydrotestosterone and an estrogen antagonist. Pharmacol Biochem Behav. 1978 Jul;9(1):81-6. doi: 10.1016/0091-3057(78)90015-1. PMID 704656
- [Background] Hayashi Y. Effects of intra-amygdaloid injections of alpha-difluoromethylornithine and putrescine on the development of electrical kindling in rats. Brain Res. 1991 Sep 27;560(1-2):181-5. doi: 10.1016/0006-8993(91)91230-x. PMID 1760726
- [Background] Shoeb M, Ramana KV. Anti-inflammatory effects of benfotiamine are mediated through the regulation of the arachidonic acid pathway in macrophages. Free Radic Biol Med. 2012 Jan 1;52(1):182-90. doi: 10.1016/j.freeradbiomed.2011.10.444. Epub 2011 Oct 24. PMID 22067901
- [Background] Newman SP. Aerosol deposition considerations in inhalation therapy. Chest. 1985 Aug;88(2 Suppl):152S-160S. doi: 10.1378/chest.88.2_supplement.152s. PMID 3893925
- [Background] Yadav UC, Kalariya NM, Srivastava SK, Ramana KV. Protective role of benfotiamine, a fat-soluble vitamin B1 analogue, in lipopolysaccharide-induced cytotoxic signals in murine macrophages. Free Radic Biol Med. 2010 May 15;48(10):1423-34. doi: 10.1016/j.freeradbiomed.2010.02.031. Epub 2010 Feb 26. PMID 20219672
- [Background] Yadav UC, Subramanyam S, Ramana KV. Prevention of endotoxin-induced uveitis in rats by benfotiamine, a lipophilic analogue of vitamin B1. Invest Ophthalmol Vis Sci. 2009 May;50(5):2276-82. doi: 10.1167/iovs.08-2816. Epub 2009 Jan 10. PMID 19136698
- [Background] Tai HH, Tong M, Ding Y. 15-hydroxyprostaglandin dehydrogenase (15-PGDH) and lung cancer. Prostaglandins Other Lipid Mediat. 2007 May;83(3):203-8. doi: 10.1016/j.prostaglandins.2007.01.007. Epub 2007 Jan 17. PMID 17481556
- [Background] Liu S, Stromberg A, Tai HH, Moscow JA. Thiamine transporter gene expression and exogenous thiamine modulate the expression of genes involved in drug and prostaglandin metabolism in breast cancer cells. Mol Cancer Res. 2004 Aug;2(8):477-87. PMID 15328374
- [Background] Rodriguez Melendez R. [Importance of water-soluble vitamins as regulatory factors of genetic expression]. Rev Invest Clin. 2002 Jan-Feb;54(1):77-83. Spanish. PMID 11995411
- [Background] Bettendorff L, Wins P. Thiamin diphosphate in biological chemistry: new aspects of thiamin metabolism, especially triphosphate derivatives acting other than as cofactors. FEBS J. 2009 Jun;276(11):2917-25. doi: 10.1111/j.1742-4658.2009.07019.x. Epub 2009 Apr 23. PMID 19490098
- [Background] Hazell AS, Butterworth RF. Update of cell damage mechanisms in thiamine deficiency: focus on oxidative stress, excitotoxicity and inflammation. Alcohol Alcohol. 2009 Mar-Apr;44(2):141-7. doi: 10.1093/alcalc/agn120. Epub 2009 Jan 16. PMID 19151161
- [Background] Desjardins P, Butterworth RF. Role of mitochondrial dysfunction and oxidative stress in the pathogenesis of selective neuronal loss in Wernicke's encephalopathy. Mol Neurobiol. 2005;31(1-3):17-25. doi: 10.1385/MN:31:1-3:017. PMID 15953809